CLINICAL TRIAL: NCT06541496
Title: Influence of Fitzpatrick Skin Phototype and Body Mass Index on Non-invasive Optoacoustic Imaging of Muscle During Vascular Restriction and Physical Activity
Brief Title: Influence of Fitzpatrick Skin Phototype and Body Mass Index on Non-invasive Optoacoustic Imaging
Status: Recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: cMSOT2-HV-01
Record Dates: First submitted 2024-06-24; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-06

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (9):
- Fitzpatrick 1: Healthy volunteers with skin type 1.
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- Fitzpatrick 2: Healthy volunteers with skin type 2.
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- Fitzpatrick 3: Healthy volunteers with skin type 3.
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- Fitzpatrick 4: Healthy volunteers with skin type 4.
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- Fitzpatrick 5: Healthy volunteers with skin type 5.
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- Fitzpatrick 6: Healthy volunteers with skin type 6.
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- BMI Group 1: Healthy volunteers with BMI <18.5.
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- BMI Group 2: Healthy volunteers with BMI >18.5 but <25.
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- BMI Group 3: Healthy volunteers with BMI >25.
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)

INTERVENTIONS:
Device: Multispectral Optoacoustic Tomography (MSOT) — Non-invasive transcutaneous MSOT imaging of muscle regions.

SUMMARY:
Multispectral Optoacoustic Tomography (MSOT) is a promising imaging technology that utilizes pulsed laser light. While melanin content in the skin has been reported to influence light-based measurements in pulse oximetry and near-infrared spectroscopy, its effects on MSOT are not well understood. This proposed study aims to investigate how different Fitzpatrick skin phenotypes (FSP) and body mass index (BMI) influence muscle perfusion and oxygenation during arterial occlusion and muscle exercise over time. Healthy volunteers with varying skin tones (as defined by FSP) and BMI will be recruited and subjected to leg arterial occlusion and toe raise exercises. They will then be scanned on different body areas (arms and legs) to assess changes in muscle perfusion and oxygenation using MSOT.

DETAILED DESCRIPTION:
Melanin, a pigment found in the skin, has been reported to influence light-based measurements such as pulse oximetry or near-infrared spectroscopy (NIRS). Studies have shown measurements overestimation of darker skin tones or in ethnicities assumed to have darker skin tones compared to lighter skin tones. Even though optoacoustic imaging (OAI) has a different depth penetration than NIRS or pulse oximetry, the technology uses pulse laser light to assess tissue.

Multispectral Optoacoustic Tomography (MSOT) imaging is similar to conventional sonography: a transducer is placed on the skin, and instead of sound, energy is applied to the tissue by means of pulsed laser light. This leads to a constant change of minimal expansion and contraction of individual tissue components or molecules. The resulting sound waves can then be detected by the same device. Previous studies have already shown that the quantitative determination of hemoglobin can provide information on inflammatory activities or muscle hemodynamics. MSOT uses laser light between 660 and 1300nm to visualize and quantify different endogenous chromophores, such as hemoglobin, collagen, or melanin. Increase in melanin concentration (e.g. in melanomas or skin tags) has been previously assessed using the technology but never looked at signal at depth. Additionally, differences in body-mass-index (BMI) might influence light penetration, and therefore, the optoacoustic signal at depth. So far, no studies have looked at the influence of increased melanin concentration or subcutaneous fat on quantification of muscle perfusion and oxygenation.

In this first pilot study, the aim is to investigate the influence of different Fitzpatrick skin phenotypes (FSP) and BMI on muscle perfusion and oxygenation during arterial occlusion or muscle exercise and over time. This information is essential for further studies with a more diverse study population.

To gain insights into these differences, healthy volunteers with different skin tone (defined by FSP) and body-mass-index will be recruited and subjected to a leg arterial occlusion and to perform a toe raise exercise. They will then be scanned on different body areas (arm, legs) to assess changes in muscle perfusion and oxygenation by MSOT.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent

Exclusion Criteria:

* Pregnancy
* diagnosed diabetes
* diagnosed renal insufficiency
* diagnosed Peripheral arterial disease
* diagnosed muscle associated disease
* tattoos in scan area
* missing consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible subjects are healthy volunteers who will be recruited from advertised announcements.
  All subjects meeting all inclusion and none of the exclusion criteria will be enrolled.
  Each healthy volunteer is categorized in 2 different groups based on his FSP and BMI:
  1. FSP I, II, III, IV, V or VI, using the filled Fitzpatrick scale self-assessment questionnaire.
  2. BMI<18.5 kg/m2, ≥ 18.5 and < 25 kg/m2 or ≥ 25 kg/m2, using the measured body weight and recorded body height.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative hemoglobin-associated signal (in arbitrary units) | immediately before and after intervention (occlusion and exercise)
  Hemoglobin signal in the measured muscle regions in all different cohorts

SECONDARY OUTCOMES:
Muscle oxygenation (in arbitrary units) | immediately before and after intervention (occlusion and exercise)
  Oxygenated hemoglobin signal in the measured muscle regions in all different cohorts
Oxygen saturation (in %) | immediately before and after intervention (occlusion and exercise)
  Proportion of oxygenated hemoglobin signal compared with total hemoglobin signal in the measured muscle regions in all different cohorts
Heart rate (in bpm) | immediately before and after intervention (occlusion and exercise)
  heart rate of the healthy volunteers
Blood pressure (in mm Hg) | immediately before and after intervention (occlusion and exercise)
  blood pressure of the healthy volunteers
Weight (in kg) | baseline
  measured by body scale
Age in years | baseline
  Participant questionnaire.
Gender: male, female, other | baseline
  Participant questionnaire.
Skin tone based on Fitzpatrick questionnaire self-assessment (type 1-6, 1 being the palest, 6 being the darkest) | baseline
  Participant questionnaire.
Dominant side | baseline
  Participant questionnaire.
Sport frequency | baseline
  Participant questionnaire.
Information on last physical exercise and caffeine and alcohol consumption | baseline
  Participant questionnaire.
Quantitative collagen, lipid, water and melanin signal (in arbitrary units) | immediately before and after intervention (occlusion and exercise)
  Signal in the measured muscle regions and the skin (melanin) in all different cohorts
Skin tone based on Fitzpatrick scale self-assessment (type 1-6, 1 being the palest, 6 being the darkest) | baseline
  color card as reference
Skin tone based on Fitzpatrick scale examiner-assessment (type 1-6, 1 being the palest, 6 being the darkest) | baseline
  color card as reference

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Knieling, PD Dr. med. habil., Principal Investigator — Department of Pediatrics and Adolescent Medicine, University Hospital Erlangen
Locations (1):
- iThera Medical Headquarters, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be transferred to iThera Medical GmbH in anonymized form. iThera Medical GmbH is authorized to further transfer the anonymized data to the American Food and Drug Administration. The study results will be published anonymously in a scientific journal. Additionally, the raw data is planned to be published by the Friedrich-Alexander-University in an open-source manner to serve as reference standard. However it will not be possible to draw conclusions about the identity of the participating individuals.